CLINICAL TRIAL: NCT05697770
Title: SODium BICarbonate for Metabolic Acidosis in the Intensive Care Unit (SODa-BIC): A Multicentre, Randomised, Double-blind Clinical Trial
Brief Title: SODium BICarbonate for Metabolic Acidosis in the ICU
Acronym: SODa-BIC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/ASN001
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Acidosis; Shock
Keywords: Sodium bicarbonate; Metabolic acidosis; Shock; Clinical trial
MeSH Terms: conditions — Acidosis; Shock | interventions — Sodium Bicarbonate; Glucose

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated in a 1:1 ratio to receive either an infusion of D5W + sodium bicarbonate, or D5W alone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An unblinded research coordinator, pharmacist or nurse not involved in data collection or bedside care will prepare the drug.
  The bedside nurse who administers the drug, other care providers, all investigators and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): Sodium bicarbonate 8.4% (1000 mEq/L) will be diluted in a D5W solution (500 mL bag). For preparation, 300 mL of D5W will be removed and 300 mL of sodium bicarbonate 8.4% added to prepare the bicarbonate solution in a total volume of 500 mL (final concentration: 600 mEq/L).
  Interventions: Drug: Sodium bicarbonate
- 5% dextrose (Active Comparator): Standard 500 mL bag of D5W.
  Interventions: Drug: 5% Dextrose

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate 8.4% will be continuously infused for a maximum of 5 hours. The infusion will start at 100 mL/hr and be kept at this rate until both pH and BE targets are achieved, following which, the infusion rate will be decreased to 25 mL/hr and kept constant at this rate until 5 hours has elapsed since the start of the infusion. At this point, the infusion will be stopped, independently, of the results of arterial blood gas analysis.
  Arms: Sodium bicarbonate
Drug: 5% Dextrose — 5% dextrose will be continuously infused for a maximum of 5 hours. The infusion will start at 100 mL/hr and be kept at this rate until both pH and BE targets are achieved, following which, the infusion rate will be decreased to 25 mL/hr and kept constant at this rate until 5 hours has elapsed since the start of the infusion. At this point, the infusion will be stopped, independently, of the results of arterial blood gas analysis.
  Arms: 5% dextrose

SUMMARY:
This trial aims to assess if, among adults in the ICU with metabolic acidosis, an infusion of sodium bicarbonate diluted in 5% dextrose, compared with an infusion of 5% dextrose, reduces Major Adverse Kidney Events within 30 days of randomization.

DETAILED DESCRIPTION:
Background: Metabolic acidosis refers to any process that elevates the concentration of hydrogen ions in the body, and is commonly encountered in critical illness. Lactic acidosis, diabetic ketoacidosis, and hyperchloremic acidosis are major examples seen in the intensive care unit (ICU). Metabolic acidosis may impair cardiac function, and sodium bicarbonate can be used to normalise blood pH. Despite being in common clinical usage, the clinical efficacy of sodium bicarbonate is still uncertain. Previous studies exploring the effects of sodium bicarbonate therapy have been limited and of variable quality.

Aim: This trial aims to assess if, among adults in the ICU with metabolic acidosis, an infusion of sodium bicarbonate diluted in 5% dextrose, compared with an infusion of 5% dextrose, reduces Major Adverse Kidney Events within 30 days of randomization.

Study Design: Phase 3, international, multicentre, double-blind, randomised clinical trial.

Participants: Adult patients (≥ 18 years old), admitted to the ICU within 48 hours, receiving a continuous infusion of a vasopressor drug to maintain a mean arterial pressure > 65 mmHg (or a mean arterial pressure target set by the treating clinician), a dedicated line (central or peripheral) is available (or is about to be made available within 1 hour after randomisation), and within two hours prior to randomisation the participant has metabolic acidosis, defined as: 1) pH < 7.30; 2) BE ≤ -4 mEq/L; and 3) PaCO2 ≤ 45 mmHg for non-intubated patients or PaCO2 ≤ 50 mmHg for non-intubated patients

Intervention: Patients will be randomly allocated in a 1:1 ratio to receive two treatments that are commonly used either an infusion of 5% dextrose (D5W) + sodium bicarbonate, or D5W alone, as a comparator. Study drug will be continuously infused targeting a pH 7.30 - 7.35 and a BE ≥ 0 mEq/L. The infusion will be maintained until this target is achieved and continued by titration thereafter for a maximum of 5 hours (to maintain target pH and base excess levels). All other aspects of care will be determined by the treating clinical team, including the use of additional fluid therapy, vasopressors, and other organ support modalities. Open-label sodium bicarbonate bolus infusion is allowed in both groups if clinically indicated.

Primary outcome: The primary outcome is the proportion of patients who meet one or more criteria for a major adverse kidney event within 30 days (MAKE 30). MAKE 30 is a composite of death, new receipt of renal-replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥ 200% of the baseline value). All components of MAKE30 will be censored at hospital discharge or 30 days after enrolment, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

All the diagnostic criteria of metabolic acidosis below have to be fulfilled within the last 2 hours before randomisation (pH, PaCO2 and BE from the same blood gas), and a vasopressor is being infused continuously at the time of randomization.

1. Adults (≥ 18 years);
2. Receiving a continuous infusion of a vasopressor to maintain mean arterial pressure > 65 mmHg (or a mean arterial pressure target set by the treating clinician);
3. A dedicated intravenous line (central or peripheral) is available (or insertion of such a line is planned within the next hour); and
4. Metabolic acidosis, defined as:

   1. pH < 7.30; and
   2. BE ≤ -4 mEq/L; and
   3. PaCO2 ≤ 45 mmHg for non-intubated patients or PaCO2 ≤ 50 mmHg for intubated patients.

Exclusion Criteria:

1. Fulfilled all eligibility criteria greater than 48 hours ago; or
2. Suspected clinically significant digestive or urinary tract loss of sodium bicarbonate (e.g., diarrhoea, ileostomy losses, renal tubular acidosis, or drainage of pancreatic or bile duct); or
3. DKA; or
4. Estimated glomerular filtration rate (eGFR) < 30 mL/min due to chronic kidney disease; or
5. Currently receiving sodium bicarbonate at the moment of randomisation (doses of sodium bicarbonate prior to randomisation are allowed); or
6. Currently receiving RRT (acute or chronic) or planned to start RRT in the next 3 hours (according to the treating clinical team); or
7. Severe dysnatraemia (serum Na ≥ 155 mEq/L or < 120 mEq/L); or
8. Hypokalaemia (serum K < 2.5 mEq/L); or
9. Pulmonary oedema with PaO2 / FiO2 < 100; or
10. Hypocalcaemia (iCa < 0.8mmol/L); or
11. Patients admitted to the ICU after a drug overdose or intoxication (including alcohol intoxication); or
12. Pregnancy or breastfeeding; or
13. Death is deemed to be inevitable as a result of the current acute illness and either the treating clinician, the patient or the substitute decision maker are not committed to full active treatment; or
14. Patients with a life expectancy < 30 days due to a chronic or underlying medical condition; or
15. Considered to be at high risk of cerebral oedema by the treating clinician (e.g. traumatic brain injury or acute brain disease); or
16. Clinician believes that being enrolled in intervention or control arm is not in the best interest of the patient; or
17. Previous enrolment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
MAKE30 score | 30 days or at hospital discharge (whichever occurs first)
  The primary outcome is MAKE30 from the date of randomisation. MAKE30 is defined as a composite of death from any cause, receipt of RRT, or persistent renal dysfunction (defined as an elevation of the creatinine level to ≥200% of baseline), all censored at hospital discharge or 30 days, whichever occurs first.

SECONDARY OUTCOMES:
30-day in-hospital mortality | 30 days or at hospital discharge (whichever occurs first)
  All-cause in-hospital mortality at day 30
Receipt of renal replacement therapy in the first 30 days | 30 days or at hospital discharge (whichever occurs first)
  Receipt of renal replacement therapy in the first 30 days
Persistent renal dysfunction | 30 days or at hospital discharge (whichever occurs first)
  Defined as an elevation of the creatinine level to ≥ 200% of baseline
Renal replacement therapy dependence at day 30 | 30 days or at hospital discharge (whichever occurs first)
  Defined by the receipt of any form of renal replacement therapy within ± 10 days of the 30-day time point following randomisation
ICU mortality | 30 days or at hospital discharge (whichever occurs first)
  All-cause ICU mortality at day 30
Hospital mortality | 90 days or at hospital discharge (whichever occurs first)
  All-cause hospital mortality at day 90
90-day in-hospital mortality | 90 days or at hospital discharge (whichever occurs first)
  All-cause mortality at day 90

OTHER OUTCOMES:
Recurrence of metabolic acidosis in the first 7 days after randomization | 7 days after randomization
  Defined as pH < 7.30, BE ≤ -4 mEq/L and PaCO2 ≤ 45 mmHg
Incidence and the maximum stage of AKI in the first 7 days after randomization | 7 days after randomization
  According to KDIGO criteria
Vasopressor-free days at day 30 | 30 days or at hospital discharge (whichever occurs first)
  Defined as 30 - days receiving a continuous infusion of vasopressor [at any time and for any duration]; non-survivors at day 30 will receive 0
Renal replacement therapy-free days at day 30 | 30 days or at hospital discharge (whichever occurs first)
  Defined as 30 - days receiving RRT; non-survivors at day 30 will receive 0
ICU-free days at day 30 | 30 days or at hospital discharge (whichever occurs first)
  Defined as 30 - ICU length of stay; non-survivors at day 30 will receive 0
Hospital-free days at day 90 | 90 days or at hospital discharge (whichever occurs first)
  Defined as 90 -hospital length of stay; non-survivors at day 90 will receive 0

CONTACTS AND LOCATIONS:
Overall Officials: Ary Serpa Neto, PhD, Principal Investigator — ANZIC RC, Monash university
Locations (53):
- Australia (40):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sutherland Hospital, Caringbah, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Queen Elizabeth II Jubilee Hospital, Coopers Plains, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hopsital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Grapmians Health, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Casey Hospital, Berwick, Victoria
  - The Victorian Heart Hospital, Clayton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - The Austin Hospital, Heidelberg, Victoria
  - Peninsula Private Hospital, Langwarrin, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Epworth, Richmond, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Bunbury Regional Hospital, Bunbury, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Centro de Estudos e de Pesquisas em Terapia Intensiva, Curitiba, Paraná, Brazil
- India (2):
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry
  - Deep Hospital, Ludhiana, Punjab
- The Jikei University Hospital, Minato, Tokyo, Japan
- New Zealand (7):
  - Auckland City Hospital (CVICU), Auckland, Auckland
  - Auckland City Hospital (DCCM), Auckland, Auckland
  - Middlemore Hospital, Auckland, Auckland
  - Christchurch Hospital, Christchurch, Christchurch
  - Dunedin Hospital, Dunedin, Dunedin
  - Waikato Hospital, Hamilton, Hamilton
  - Wellington Regional Hospital, Wellington
- Sultan Qaboos Comprehensive Cancer Care and Research Center, Seeb, Oman
- King Abdullah International Medical Research Center, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serpa Neto A, McNamara M, Cooper J, Fujii T, Higgins A, Hodgson C, Navarra L, Nichol A, Peake S, Rea-Neto A, Secombe P, See E, Taylor P, Young M, Zampieri FG, Young P, Bellomo R, Udy A; SODa-BIC investigators. Protocol summary and statistical analysis plan for the sodium bicarbonate for metabolic acidosis in the intensive care unit (SODa-BIC) trial. Crit Care Resusc. 2025 May 15;27(2):100108. doi: 10.1016/j.ccrj.2025.100108. eCollection 2025 Jun. PMID 40487345